CLINICAL TRIAL: NCT00724971
Title: A Phase 1 Study Of Cmc-544 Administered In Combination With Rituximab In Subjects With B-cell Non-hodgkin's Lymphoma
Brief Title: Study Evaluating The Safety And Tolerability Of Combination Therapy Inotuzumab Ozogamicin (CMC-544) And Rituximab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3129K3-1104; B1931005 (Other: Alias Study Number)
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Lymphoma, B-Cell
Keywords: B-cell Non-Hodgkin's Lymphoma; NHL
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Inotuzumab Ozogamicin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inotuzumab Ozogamicin + Rituximab (Experimental)
  Interventions: Drug: Inotuzumab Ozogamicin (CMC-544); Drug: Rituximab (Rituxan)

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin (CMC-544) — 1.8 mg/m2, IV on day 2 of each 28 day cycle; up to 8 cycles unless PD, unacceptable toxicity, or subject's refusal occurs.
Drug: Rituximab (Rituxan) — 375 mg/m2, IV on day 1 of each 28 day cycle; up to 8 cycles unless PD, unacceptable toxicity, or subject's refusal occurs.

SUMMARY:
To assess the tolerability and the initial safety profile of Inotuzumab Ozogamicin (CMC-544) in combination with Rituximab in patients with B-Cell Non-Hodgkin's lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria:

* CD20 and CD22-positive, B-cell NHL which has progressed after 1 or 2 prior therapies.
* Prior therapy must have contained at least one dose of Rituximab therapy. Patients can not be refractory to Rituximab (refractory = PD under treatment or within 6 month
* Eastern Cooperative Oncology Group (ECOG) performance status: 0/ 1.
* Patients must not have received previous radioimmunotherapy.
* Patients tolerant to Rituximab.
* Patients must not have received chemotherapy, cancer immunosuppressive therapy, growth factors (except erythropoietin), or investigational agents within 28 days before first dose of test article.

Exclusion Criteria:

* Candidate for potentially curative therapies
* Subjects must not have received previous radioimmunotherapy.
* Subjects with autologous hematopoietic stem cell transplant within the last 6 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07-04 (Actual); Primary Completion 2010-03-10 (Actual); Study Completion 2010-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Japan (4):
  - Nagoya Daini Red Cross Hospital, Aichi
  - Tokai University Hospital, Kanagawa
  - National Cancer Center Hospital, Tokyo
  - Cancer Inst. Hp. of Japanese Foundation for Cancer Research, Tokyo

REFERENCES:
- [Derived] Ogura M, Hatake K, Ando K, Tobinai K, Tokushige K, Ono C, Ishibashi T, Vandendries E. Phase I study of anti-CD22 immunoconjugate inotuzumab ozogamicin plus rituximab in relapsed/refractory B-cell non-Hodgkin lymphoma. Cancer Sci. 2012 May;103(5):933-8. doi: 10.1111/j.1349-7006.2012.02241.x. Epub 2012 Mar 20. PMID 22335424
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3129K3-1104&StudyName=Study%20Evaluating%20The%20Safety%20And%20Tolerability%20Of%20Combination%20Therapy%20Inotuzumab%20Ozogamicin%20%28CMC-544%29%20And%20Rituximab

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six consecutive patients were enrolled as the first cohort. The dose and administration were considered to be reasonable if <=2 participants in the first cohort experienced a dose limiting toxicity (DLT), and an additional 4 subjects were to be enrolled as the expanded cohort for a total 10 participants.
Groups:
- CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2: Participants were treated with intravenous rituximab (375 mg/m^2) followed by intravenous CMC-544 (1.8 mg/m^2) every 28 days (±2 days) for 4 cycles (1 cycle = 28 days), and participants with at least "stable disease (SD)" after the fourth cycle received CMC-544 up to 8 cycles unless they experienced progressive disease (PD) or an unacceptable toxicity, or withdrew consent.
Period: Overall Study
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Started | 10
Completed | 4
Not Completed | 6
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.20 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: A DLT was defined as the following drug-related adverse event which occurred during the first 28 days: 1) Any National Cancer Institute (NCI) Grade 3 or 4 nonhematologic toxicity (except Grade 3 nausea or vomiting without optimal treatment), 2) Febrile neutropenia, 3) Grade 4 absolute neutrophil count lasting >=7 days, 4) Grade 4 thrombocytopenia lasting >=3 days, 5) Grade 3 or 4 thrombocytopenia associated with a bleeding episode requiring platelet transfusion, 6)Delayed recovery (to grade <=1 or baseline, except alopecia) from a drug-related toxicity that delayed the next dose >2 weeks
Time Frame: Up to 28 days
Population: The first cohort was analyzed for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 6
Participants | 2

2. Secondary Outcome: Number of Participants With Objective Response: Evaluable Population
Description: Number of participants with objective response of complete response (CR), complete response unconfirmed (CRu), or partial response (PR). Objective response included subjects with CR, CRu, and PR. Response criteria for Non-Hodgkin's Lymphoma (NHL) were based on the 1999 NCI International Workshop to standardize response criteria for NHL. Per the criteria for Lymph node masses: CR, normal size; CRu, normal or >75% decrease in the sum of the products of the greatest diameters (SPD); PR, normal or >=50% decrease in the SPD.
Time Frame: Up to 8 cycles (1 cycle = 28 days)
Population: The evaluable population included all participants who received at least 2 doses of the test article and who had a baseline tumor CT scan and underwent at least 1 postbaseline tumor assessment for anticancer clinical activity.
Measure: Count of Participants; unit: Participants
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8
Participants
  Complete response (CR) | 6
  Complete response unconfirmed (CRu) | 1
  Partial response (PR) | 0
  Objective Response (CR+CRu+PR) | 7

3. Secondary Outcome: Number of Participants With Objective Response: Intent-to-treat (ITT) Population
Description: as for outcome 2
Time Frame: Up to 8 cycles (1 cycle = 28 days)
Population: The ITT population included all participants who were enrolled in the intended dose scheme.
Measure: Count of Participants; unit: Participants
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10
Participants
  Complete response (CR) | 6
  Complete response unconfirmed (CRu) | 1
  Partial response (PR) | 1
  Objective Response (CR+CRu+PR) | 8

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: The interval from the date of first administration of the test article until the first date on which relapsed disease, progressive disease (PD), or death was documented, censored at the last tumor evaluation date. Response criteria for Non-Hodgkin's Lymphoma (NHL) were based on the 1999 NCI International Workshop to standardize response criteria for NHL. Per the criteria for Lymph node masses: Relapse/PD, appearance of any new lesion or increased by >=50% in the size.
Time Frame: Up to 591 days
Population: The evaluable population included all participants who received at least 2 doses of the test article and who had a baseline tumor computed tomography (CT) scan and underwent at least 1 postbaseline tumor assessment for anticancer clinical activity.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8
weeks | NA [NA to NA] — The number of event (PD or death) was not sufficient to estimate the median PFS.

5. Other Pre Specified Outcome: Maximum Observed Serum Concentration (Cmax) of CMC-544, Total Calicheamicin, and Anti-human CD22 Antibody (G544)
Description: CMC-544 is composed of G544, an anti-human CD22 antibody, linked to a potent cytotoxic antitumor antibiotic called calicheamicin. CD22 is expressed on the malignant cells of the majority of B-lymphocyte malignancies.
Time Frame: Cycle 1, Cycle 2 and Cycle 3 at hour 0 (predose) and at hours 1 (before the end of infusion), 4, 48, 144,192, 312, 480, and 648 relative to the start of infusion of CMC-544
Population: Phamacokinetic population included participants who received at least 1 dose of the test article and with serum concentrations available. Number Analyzed = number of participants with the pertinent parameters calculated at the visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10
ng/mL
  CMC-544: Cycle 1 | 559 (136)
  CMC-544: Cycle 2: number analyzed (Participants) | 5
  CMC-544: Cycle 2 | 822 (152)
  CMC-544: Cycle 3: number analyzed (Participants) | 3
  CMC-544: Cycle 3 | 958 (64.0)
  Total Calicheamicin: Cycle 1 | 67.7 (14.9)
  Total Calicheamicin: Cycle 2: number analyzed (Participants) | 5
  Total Calicheamicin: Cycle 2 | 80.2 (11.3)
  Total Calicheamicin: Cycle 3: number analyzed (Participants) | 3
  Total Calicheamicin: Cycle 3 | 96.6 (2.89)
  G544: Cycle 1 | 839 (157)
  G544: Cycle 2: number analyzed (Participants) | 5
  G544: Cycle 2 | 1110 (88.9)
  G544: Cycle 3: number analyzed (Participants) | 3
  G544: Cycle 3 | 1210 (177)

6. Other Pre Specified Outcome: Serum Decay Half-Life (t1/2) of CMC-544, Total Calicheamicin, and G544
Description: The time measured for the serum concentration to decrease by one half.
Time Frame: as for outcome 5
Population: Pharmacokinetic population included participants who received at least 1 dose of the test article and with serum concentrations available. Number Analyzed = number of participants with the pertinent parameters calculated at the visit.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10
hours
  CMC-544: Cycle 1: number analyzed (Participants) | 2
  CMC-544: Cycle 1 | 18.77 (1.09)
  CMC-544: Cycle 2: number analyzed (Participants) | 2
  CMC-544: Cycle 2 | 29.08 (21.79)
  CMC-544: Cycle 3: number analyzed (Participants) | 3
  CMC-544: Cycle 3 | 51.70 (20.59)
  Total Calicheamicin: Cycle 1: number analyzed (Participants) | 7
  Total Calicheamicin: Cycle 1 | 61.23 (34.84)
  Total Calicheamicin: Cycle 2: number analyzed (Participants) | 5
  Total Calicheamicin: Cycle 2 | 96.44 (31.31)
  Total Calicheamicin: Cycle 3: number analyzed (Participants) | 3
  Total Calicheamicin: Cycle 3 | 167.87 (72.85)
  G544: Cycle 1: number analyzed (Participants) | 9
  G544: Cycle 1 | 67.14 (31.84)
  G544: Cycle 2: number analyzed (Participants) | 5
  G544: Cycle 2 | 101.59 (34.08)
  G544: Cycle 3: number analyzed (Participants) | 3
  G544: Cycle 3 | 127.57 (32.76)

7. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of CMC-544, Total Calicheamicin, and G544
Description: AUClast= Area under the serum concentration versus time curve from time zero (pre-dose) to time of last measured concentration.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10
ng*hour/mL
  CMC-544: Cycle 1 | 12300 (6200)
  CMC-544: Cycle 2: number analyzed (Participants) | 5
  CMC-544: Cycle 2 | 27000 (7450)
  CMC-544: Cycle 3: number analyzed (Participants) | 3
  CMC-544: Cycle 3 | 50100 (6390)
  Total Calicheamicin: Cycle 1 | 2850 (1400)
  Total Calicheamicin: Cycle 2: number analyzed (Participants) | 5
  Total Calicheamicin: Cycle 2 | 6490 (2250)
  Total Calicheamicin: Cycle 3: number analyzed (Participants) | 3
  Total Calicheamicin: Cycle 3 | 10700 (4750)
  G544: Cycle 1 | 38400 (16300)
  G544: Cycle 2: number analyzed (Participants) | 5
  G544: Cycle 2 | 84900 (23400)
  G544: Cycle 3: number analyzed (Participants) | 3
  G544: Cycle 3 | 127000 (44800)

8. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC∞) of CMC-544, Total Calicheamicin, and G544
Description: AUC∞ = Area under the serum concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10
ng*hour/mL
  CMC-544: Cycle 1: number analyzed (Participants) | 2
  CMC-544: Cycle 1 | 22300 (2850)
  CMC-544: Cycle 2: number analyzed (Participants) | 2
  CMC-544: Cycle 2 | 34800 (12200)
  CMC-544: Cycle 3: number analyzed (Participants) | 3
  CMC-544: Cycle 3 | 54800 (7070)
  Total Calicheamicin: Cycle 1: number analyzed (Participants) | 7
  Total Calicheamicin: Cycle 1 | 4060 (1100)
  Total Calicheamicin: Cycle 2: number analyzed (Participants) | 5
  Total Calicheamicin: Cycle 2 | 7460 (2540)
  Total Calicheamicin: Cycle 3: number analyzed (Participants) | 3
  Total Calicheamicin: Cycle 3 | 12700 (5400)
  G544: Cycle 1: number analyzed (Participants) | 9
  G544: Cycle 1 | 47700 (14300)
  G544: Cycle 2: number analyzed (Participants) | 5
  G544: Cycle 2 | 92300 (26300)
  G544: Cycle 3: number analyzed (Participants) | 3
  G544: Cycle 3 | 138000 (42600)

9. Other Pre Specified Outcome: Clearance (CL) of CMC-544, Total Calicheamicin, and G544
Description: The rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10
L/hour
  CMC-544: Cycle 1: number analyzed (Participants) | 2
  CMC-544: Cycle 1 | 0.120 (0.0185)
  CMC-544: Cycle 2: number analyzed (Participants) | 2
  CMC-544: Cycle 2 | 0.0782 (0.0192)
  CMC-544: Cycle 3: number analyzed (Participants) | 3
  CMC-544: Cycle 3 | 0.0499 (0.0012)
  Total Calicheamicin: Cycle 1: number analyzed (Participants) | 7
  Total Calicheamicin: Cycle 1 | 0.746 (0.212)
  Total Calicheamicin: Cycle 2: number analyzed (Participants) | 5
  Total Calicheamicin: Cycle 2 | 0.424 (0.133)
  Total Calicheamicin: Cycle 3: number analyzed (Participants) | 3
  Total Calicheamicin: Cycle 3 | 0.249 (0.0686)
  G544: Cycle 1: number analyzed (Participants) | 9
  G544: Cycle 1 | 0.0662 (0.0236)
  G544: Cycle 2: number analyzed (Participants) | 5
  G544: Cycle 2 | 0.0331 (0.0077)
  G544: Cycle 3: number analyzed (Participants) | 3
  G544: Cycle 3 | 0.0213 (0.0062)

10. Other Pre Specified Outcome: Volume of Distribution (Vss) of CMC-544, Total Calicheamicin, and G544
Description: The theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10
L
  CMC-544: Cycle 1: number analyzed (Participants) | 2
  CMC-544: Cycle 1 | 2.33 (0.0763)
  CMC-544: Cycle 2: number analyzed (Participants) | 2
  CMC-544: Cycle 2 | 2.26 (1.74)
  CMC-544: Cycle 3: number analyzed (Participants) | 3
  CMC-544: Cycle 3 | 3.02 (1.23)
  Total Calicheamicin: Cycle 1: number analyzed (Participants) | 7
  Total Calicheamicin: Cycle 1 | 47.6 (11.3)
  Total Calicheamicin: Cycle 2: number analyzed (Participants) | 5
  Total Calicheamicin: Cycle 2 | 45.6 (7.04)
  Total Calicheamicin: Cycle 3: number analyzed (Participants) | 3
  Total Calicheamicin: Cycle 3 | 47.8 (6.62)
  G544: Cycle 1: number analyzed (Participants) | 9
  G544: Cycle 1 | 3.95 (0.921)
  G544: Cycle 2: number analyzed (Participants) | 5
  G544: Cycle 2 | 3.39 (0.515)
  G544: Cycle 3: number analyzed (Participants) | 3
  G544: Cycle 3 | 3.02 (0.400)

11. Other Pre Specified Outcome: Number of Participants With Positive Serum Antibody to Inotuzumab Ozogamicin (CMC-544)
Description: Antibody responses to CMC-544
Time Frame: Up to 8 Cycles (1 cycle = 28 days)
Population: The intent-to-treat (ITT) population included all participants in the intended dose scheme.
Measure: Count of Participants; unit: Participants
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10
Participants
  Screening | 1
  End of Treatment | 0

12. Other Pre Specified Outcome: Number of Participants With Positive Serum Antibody to Rituximab
Description: Antibody responses to rituximab
Time Frame: Up to 8 Cycles (1 cycle = 28 days)
Population: The intent-to-treat (ITT) population included all participants in the intended dose scheme.
Measure: Count of Participants; unit: Participants
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10
Participants
  Screening | 0
  End of Treatment | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CMC-544 1.8 mg/m^2 + Rituximab 375 mg/m^2 (N=10)
Anaemia (Blood and lymphatic system disorders) | 1
Erythropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 8
Lymphocytosis (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 6
Monocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Arrhythmia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Extravasation (General disorders) | 1
Fatigue (General disorders) | 5
Influenza like illness (General disorders) | 1
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 2
Pyrexia (General disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 4
Cytokine release syndrome (Immune system disorders) | 1
Food allergy (Immune system disorders) | 1
Cystitis bacterial (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Mouth injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 9
Blood alkaline phosphatase increased (Investigations) | 5
Blood amylase increased (Investigations) | 1
Blood calcium increased (Investigations) | 1
Blood glucose increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 6
Blood potassium decreased (Investigations) | 1
Blood sodium increased (Investigations) | 1
C-reactive protein increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 3
Glucose urine present (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 3
Protein total decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Monarthritis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Lethargy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.